CLINICAL TRIAL: NCT00298805
Title: Dysphoric-like Disorder of Epilepsy, Is It Unique?
Brief Title: A Quality of Life Study in Patients With Migraines
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to expiration of IRB approval
Sponsor: Northwell Health (Other)
Collaborators: Rush University Medical Center (Other); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 05.02.073
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Migraine; Headache; Depression
Keywords: Migraine; Headache; Depression; Quality of Life
MeSH Terms: conditions — Migraine Disorders; Headache; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare depressive characteristics in migraine patients to those observed in patients with epilepsy in a previous study, and determine whether those symptoms are unique to patients with epilepsy.

DETAILED DESCRIPTION:
A form of depression known as dysphoric-like disorder is common in people with epilepsy, which may significantly affect the quality of life in these people, as shown in a previous study. However, it is unclear if this depressive disorder is unique to patients with epilepsy. In order to assess whether these symptoms are unique and idiosyncratic to the epilepsy population, in this multi-center study, these dysphoric depressive features will be contrasted to those seen in patients with other neurologic or psychiatric conditions. Migraine is selected as one of the comparison disorders because it shares with epilepsy characteristics of being a recurrent episodic central nervous system disorder, and our site will only enroll patients with migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Have the diagnosis of migraine
* Have had no change in migraine medication(s) 30 days prior to study
* Achieve a satisfactory score on the Wide Range Achievement Test 3 (WRAT3) test at the screening visit
* Capable of completing self-reporting questionnaires
* Willing and able to provide written informed consent and comply with the study protocol

Exclusion Criteria:

* Presence of a clinically significant comorbidity of an unstable or progressive nature
* Presence of major depression
* Participation in an investigational drug study within the past 30 days
* Inability to communicate well with site study personnel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Migraine patients will be recruited from the outpatient neurology clinics / offices.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2006-01; Primary Completion 2009-06 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Dysphoric-like depressive characteristics in patient with epilepsy | N/A (cross-sectional study)

CONTACTS AND LOCATIONS:
Overall Officials: Andres M Kanner, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- North Shore Long Island Jewish Health System, Great Neck, New York, United States